CLINICAL TRIAL: NCT02116751
Title: Frequency and Clinical Significance of Renal and Bone Toxicity in HIV-infected Patients: Role of Classical Factors, HIV Infection, and Antiretroviral Therapy
Brief Title: Frequency and Clinical Significance of Renal and Bone Toxicity in HIV-infected Patients
Acronym: ComorVIH
Status: Completed | Type: Observational
Sponsor: Asociacion para el Estudio de las Enfermedades Infecciosas (Network)
Responsible Party: Sponsor
Other Study IDs: EC 039/14
Record Dates: First submitted 2014-04-11; First posted 2014-04-17 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-04

CONDITIONS: Renal Toxicity
Keywords: HIV, antiretroviral, toxicity, eGFR, tubular disease, BMD

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine the frequency of renal and bone toxicity in HIV infected patients receiving antiretroviral therapy, and the outcome in terms of treatment change or/and virological failure, in relation with the presence of classical factors, such as diabetes or hypertension, the role of HIV itself, because of chronic inflammation, and the effects of antiretroviral medication.

DETAILED DESCRIPTION:
This is a retrospective cohort study involving 300 patients to determine the frequency of renal and bone comorbidities/toxicity in a large population of HIV-infected patients receiving antiretroviral therapy, in order to establish the differential role of classical factors, HIV infection, or antiretroviral therapy.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed HIV infection

Exclusion Criteria:

* Pregnancy
* Prior therapy with antineoplastic chemotherapy or chronic treatment with corticosteroids
* Previous chronic therapy with antiresorptive bone therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV infected patients in active follow up, receiving antiretroviral therapy
Sampling Method: Non-Probability Sample
Enrollment: 306 (Actual)
Dates: Start 2014-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Incidence of Renal and Bone toxicity | Patients will be evaluated for 2 years before
  Number and percentage of patients with:
  * Confirmed estimated glomerular filtration rate (eGFR) by CKD (chronic kidney disease)-epi equation decrease to < 60 ml/min, or/and
  * More than 25% of eGFR decrease during therapy, or/and
  * Tubular toxicity defined as at least two of confirmed proteinuria (> 300 mg/g), glycosuria with euglycemia, fractional excretion of urinary phosphate > 20%, or of uric acid > 10%. AND
  * Number and percentage of patients with bone mineral density (BMD) decrease > 10% during follow up or progression to osteopenia (from normal) or to osteoporosis (from osteopenia)

SECONDARY OUTCOMES:
Consequences of renal or bone toxicity | Patients will be evaluated for 2 years before
  Percentage of patients with regimen discontinuation (any drug in the regimen) because of renal or/and bone toxicity

OTHER OUTCOMES:
Changes in renal and bone toxicity | 2 years before entry
  Evolution of renal and bone parameters in case of regimen discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Jose L Casado, MD, Principal Investigator — Ramon y Cajal Hospital
Locations (1):
- Ramon y Cajal Hospital, Madrid, Madrid, Spain